CLINICAL TRIAL: NCT06605599
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Fixed-dose Study to Evaluate the Efficacy, Safety, and Tolerability of ABBV-932 in Subjects With Depressive Episodes Associated With Bipolar I or II Disorder
Brief Title: Study of Oral ABBV-932 to Assess Adverse Events and Change in Disease Activity in Adult Participants With Bipolar I or II Disorder
Acronym: CANTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-894
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Bipolar I Disorder; Bipolar II Disorder
Keywords: Bipolar I Disorder; Bipolar II Disorder; Bipolar Disorder; ABBV-932
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- ABBV-932 Dose A (Experimental): Participants will receive ABBV-932 Dose A.
  Interventions: Drug: ABBV-932
- ABBV-932 Dose B (Experimental): Participants will receive ABBV-932 Dose B.
  Interventions: Drug: ABBV-932
- ABBV-932 Dose C (Experimental): Participants will receive ABBV-932 Dose C.
  Interventions: Drug: ABBV-932
- Placebo for ABBV-932 (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo for ABBV-932

INTERVENTIONS:
Drug: ABBV-932 — Oral Capsule
  Arms: ABBV-932 Dose A; ABBV-932 Dose B; ABBV-932 Dose C
Drug: Placebo for ABBV-932 — Oral Capsule
  Arms: Placebo for ABBV-932

SUMMARY:
Bipolar disorder is a severe chronic mood disorder that affects up to 4% of the adult population in the United States. This study will assess how safe and effective ABBV-932 is in treating participants with bipolar I or II disorder.

ABBV-932 is an investigational drug being developed for the treatment of depressive episodes in adult participants with bipolar I or II disorder. Study doctors put participants in 1 of 4 groups, called treatment arms. There is a 1 in 4 chance that a participant will be assigned to placebo. Around 160 adult participants with bipolar I or II disorder will be enrolled in approximately 40 sites worldwide.

Participants will receive oral capsules of ABBV-932 or matching placebo once daily for 6 weeks. The treatment period will be followed by a safety follow-up (SFU) period for 4 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular weekly visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) criteria for bipolar I or II disorder without psychotic features based on the Mini International Neuropsychiatric Interview (MINI), with a current depressive episode of at least 4 weeks and not exceeding 12 months.
* Have a minimum score of 20 on the 17-item Hamilton Depression Rating Scale (HAMD-17).
* Have a minimum score of 2 on Item 1 of the HAMD-17 at screening.

Exclusion Criteria:

* Positive urine drug screen (UDS) result at screening.
* Treated with any investigational drug within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug, is currently enrolled in another clinical study, or was previously enrolled in this study.
* Current use of any antipsychotic, antidepressant, anticonvulsant, mood stabilizer, herb, or over-the-counter medication with psychoactive potential within 1 week or 5 half-lives of the medication (whichever is longer).
* Prior exposure to ABBV-932 within 90 days prior to baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score | Up to Week 6
  The MADRS is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology. Each item is scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity.

SECONDARY OUTCOMES:
Change From Baseline in Clinical Global Impression-Severity - Bipolar Disorder (CGI-S-BP) | Up to Week 6
  CGI-S-BP is a single-item clinician-reported measure of severity of bipolar disorder. Clinicians are asked to rate the severity of mania, depression, and overall bipolar illness. Response options range from 1 to 7: 1 = normal, not ill through 7 = very severely ill.
Change From Baseline in Functioning Assessment Short Test (FAST) Total Score | Up to Week 6
  FAST is a clinician-reported outcome measure designed to assess the main functioning problems experienced by psychiatric participants, particularly bipolar participants. The FAST includes 24 items in 6 domains of functioning. Clinicians are asked to respond on a 4-point Likert scale ranging from 0 to 3 (0 = no difficulty and 3 = severe difficulty). Higher scores indicate greater difficulties in functioning.
Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score | Up to Week 6
  HAM-A is a 14-item, clinician-reported measure used to quantify and categorize the participant's anxiety over the past week. Items are rated on a 5-point Likert rating scale of "absent" (0; if symptoms are absent, insignificant, or clearly due to causes other than anxiety) through "very severe" (4; if symptom is incapacitating). The HAM-A total score ranges from 0 to 56, with higher scores indicating greater anxiety severity.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (40):
- United States (32):
  - Harmonex /ID# 267504, Dothan, Alabama
  - Advanced Research Center /ID# 267716, Anaheim, California
  - Axiom Research /ID# 267518, Colton, California
  - Collaborative Neuroscience Research - Garden Grove /ID# 267654, Garden Grove, California
  - Sun Valley Research Center /ID# 267708, Imperial, California
  - Alliance for Research Alliance for Wellness /ID# 267492, Long Beach, California
  - Excell Research /ID# 267541, Oceanside, California
  - Viking Clinical Research Center - Temecula /ID# 267634, Temecula, California
  - Accel Research Sites Network - St. Pete /ID# 267463, Largo, Florida
  - GMI Florida - Central Miami Medical Institute /ID# 267566, Miami, Florida
  - Allied Biomedical Res Inst Inc /ID# 267481, Miami, Florida
  - K2 Medical Research - Orlando - South Orlando Avenue /ID# 267567, Orlando, Florida
  - Segal Trials - West Broward Outpatient Research Site /ID# 267947, Tamarac, Florida
  - Benchmark Research /ID# 267626, Shreveport, Louisiana
  - CenExel /ID# 267675, Gaithersburg, Maryland
  - Arch Clinical Trials /ID# 267507, St Louis, Missouri
  - Duplicate_Oasis Clinical Research, LLC /ID# 267969, Las Vegas, Nevada
  - Center For Emotional Fitness - Cherry Hill /ID# 267661, Cherry Hill, New Jersey
  - Bio Behavioral Health /ID# 267493, Toms River, New Jersey
  - Neurobehavioral Research /ID# 267564, Cedarhurst, New York
  - New Hope Clinical Research - Inpatient unit /ID# 267465, Charlotte, North Carolina
  - Quest Therapeutics of Avon Lake /ID# 267558, Avon Lake, Ohio
  - OSU Psychiatry Department /ID# 267730, Columbus, Ohio
  - Sooner Clinical Research /ID# 267639, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research /ID# 267451, Allentown, Pennsylvania
  - Suburban Research Associates - Media /ID# 267621, Media, Pennsylvania
  - Coastal Carolina Research Center, LLC /ID# 267550, Charleston, South Carolina
  - FutureSearch Trials of Dallas /ID# 267715, Dallas, Texas
  - Perceptive Pharma Research /ID# 267563, Richmond, Texas
  - Grayline Research Center /ID# 267466, Wichita Falls, Texas
  - Northwest Clinical Research Center /ID# 267505, Bellevue, Washington
  - Core Clinical Research /ID# 268534, Everett, Washington
- Japan (5):
  - Kokura Mental Clinic /ID# 268031, Kitakyushu, Fukuoka
  - Kawamura Mental Clinic /ID# 268325, Sapporo, Hokkaido
  - Yutaka Clinic /ID# 268026, Sagamihara, Kanagawa
  - Kaku Mental Clinic /ID# 268020, Fukuoka
  - Kuramitsu Hospital /ID# 268751, Fukuoka
- Puerto Rico (3):
  - INSPIRA Clinical Research /ID# 267041, San Juan
  - Instituto De Neurologia Dra. Ivonne Fraga, Psc /ID# 267065, San Juan
  - BDH Research /ID# 267025, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-894